CLINICAL TRIAL: NCT00404586
Title: A Randomised, Placebo-controlled, 4-period, Incomplete Block, Crossover Study of 7 Days Dosing of Intranasal GW784568X (100mcg, 200mcg and 400mcg od), Fluticasone Propionate (200mcg od) and Placebo (Blinded for GW784568X vs Placebo) to Evaluate the Efficacy and Safety Using an Environmental Chamber in Male Subjects With Allergic Rhinitis
Brief Title: Effects Of Single Doses Of GW784568X On Allergic Rhinitis Symptoms In Male Subjects Whilst In An Environmental Chamber
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: BGS105049
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Environmental Challenge Chamber; GW784568X; Intranasal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment period 1 (Experimental): In treatment period subjects will receive once daily 100 mcg of GW784568X and fluticasone propionate 200 mcg once daily for 7 days. Subjects will receive GW784568X and fluticasone propionate via intranasal route. There will be a wash out period of 14 days.
  Interventions: Drug: GW784568X; Drug: Fluticasone propionate
- Treatment period 2 (Experimental): In treatment period subjects will receive once daily 200 mcg of GW784568X and fluticasone propionate 200 mcg once daily for 7 days. Subjects will receive GW784568X and fluticasone propionate via intranasal route. There will be a wash out period of 14 days.
  Interventions: Drug: GW784568X; Drug: Fluticasone propionate
- Treatment period 3 (Experimental): In treatment period subjects will receive once daily 400 mcg of GW784568X and fluticasone propionate 200 mcg once daily for 7 days. Subjects will receive GW784568X and fluticasone propionate via intranasal route. There will be a wash out period of 14 days.
  Interventions: Drug: GW784568X; Drug: Fluticasone propionate
- Treatment period 4 (Placebo Comparator): In treatment period subjects will receive once daily Placebo and fluticasone propionate 200 mcg once daily for 7 days. Subjects will receive Placebo and fluticasone propionate via intranasal route. There will be a wash out period of 14 days.
  Interventions: Drug: Fluticasone propionate; Drug: Placebo

INTERVENTIONS:
Drug: GW784568X — GW784568X will be delivered as a micronized suspension (50 or 100mcg/spray) via an aqueous nasal spray. Dose planned for treatment groups are 100, 200 and 400 mcg.
  Arms: Treatment period 1; Treatment period 2; Treatment period 3
Drug: Fluticasone propionate — Fluticasone propionate will be delivered 50 mcg/spray and planned dose is 200 mcg.
Drug: Placebo — Matching Placebo to GW784568X as aqueous nasal spray.
  Arms: Treatment period 4

SUMMARY:
This study was designed to look at safety aspects and effects of intranasal doses of GW784568X on allergic rhinitis symptoms to develop this drug for its use in people who suffer with allergic rhinitis

DETAILED DESCRIPTION:
A randomised, placebo-controlled, 4-period, incomplete block, crossover study of 7 days dosing of intranasal GW784568X (100mcg, 200mcg and 400mcg od), fluticasone propionate (200mcg od) and placebo (blinded for GW784568X vs placebo) to evaluate the efficacy and safety using an environmental chamber in male subjects with allergic rhinitis

ELIGIBILITY:
Inclusion criteria:

* Healthy with exception of seasonal rhinitis. May also have mild asthma.
* Weight greater than or equal to 50kg
* Non-smoker for at least 12 months

Exclusion criteria:

* History of frequent nosebleeds
* Have participated in another trial in the last 30 days.
* Have donated blood in the previous 3 months
* Have used prescription or non prescription drugs within last 7 days
* Have history of alcohol/drug abuse within last 12 months
* Have positive Hepatitis B or C test within 3 months of screening
* Subject tested positive for HIV

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-09-11 (Actual); Primary Completion 2007-01-16 (Actual); Study Completion 2007-01-16 (Actual)

PRIMARY OUTCOMES:
Nasal symptom scores after 7 days of dosing | after 7 days of dosing

SECONDARY OUTCOMES:
Nasal symptom scores Eye symptom scores Other symptom scores Nasal secretion and airflow on Day 7 and Day 8 after being exposed to allergen | on Day 7 and Day 8

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany

REFERENCES:
- See also: Results for study BGS105049 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/BGS105049?search=study&search_terms=BGS105049#rs